CLINICAL TRIAL: NCT03067402
Title: Routine Or Selective Stress Testing After Revascularization: ROSSTAR Trial RCT Outline
Acronym: ROSSTAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Dominique Joyal, Interventional Cardiologist, Assistant Professor of Medicine, McGill University, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CODIM-MBM-17-001
Record Dates: First submitted 2017-02-24; First posted 2017-03-01 (Actual); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Coronary Heart Disease; Coronary Artery Disease
Keywords: Myocardial Infarction; Physiological Stress Test; Nuclear Image Perfusion; Angioplasty; Coronary Artery Bypass Graft; Percutaneous Coronary Intervention; Angina; Ischemia
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Myocardial Infarction; Angina Pectoris; Ischemia | interventions — Observation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observation (Other): Patient receives standard observation, i.e. only do a nuclear imaging stress test if symptoms present themselves over the course of 3 years.
  Interventions: Other: Observation
- Nuclear Perfusion Imaging Stress Test (Experimental): Patient receives routine nuclear image perfusion stress test
  Interventions: Diagnostic Test: Nuclear Perfusion Imaging Stress Test

INTERVENTIONS:
Other: Observation — Patient receives standard observation i.e. only do a nuclear imaging stress test if symptoms present themselves over the course of 3 years
  Arms: Observation
Diagnostic Test: Nuclear Perfusion Imaging Stress Test — Patient receives routine nuclear image perfusion stress test
  Arms: Nuclear Perfusion Imaging Stress Test

SUMMARY:
The ROSSTAR trial is a pragmatic trial that will directly compare the strategies of routine and selective stress imaging testing (with radionuclide imaging (RNI)) late after PCI or CABG in asymptomatic patients. The study will be a single center trial based at the Jewish General Hospital (JGH), a McGill University teaching hospital (Montreal, Quebec). A total of 1100 patients who are either >5 years post-CABG or >2 years post-PCI will be randomized. Half of the patients will be randomized to a routine RNI testing, and the other half to selective RNI testing.

DETAILED DESCRIPTION:
There is no consensus in current guidelines regarding the role of stress imaging testing late after revascularization. The issue to be resolved by the trial is whether routine stress imaging testing (stress test with nuclear perfusion imaging) benefits patients late after percutaneous coronary intervention (PCI) or coronary artery bypass graft surgery (CABG).

What are the principal research questions to be addressed?

1. Is a strategy of routine stress imaging testing late after PCI or CABG associated with lower clinical event rates than a strategy of selective stress imaging testing?
2. Is a strategy of routine stress imaging testing late after PCI or CABG associated with better quality of life than a strategy of selective stress imaging testing?
3. What are the resources utilization associated with routine vs. selective stress imaging testing?

What is the primary hypothesis? The primary hypothesis is that routine stress imaging testing late after PCI or CABG is associated with lower clinical event rates than a strategy of selective stress imaging testing.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients who have undergone CABG or PCI.
* 2.CABG surgery occurred >5 years and PCI >2 years prior to randomization.
* 3.Patients must have had at least one SVG in the CABG group.
* 4.Patients are asymptomatic or have minimal chronic anginal symptoms.

Exclusion Criteria:

* 1.Participation in a conflicting clinical study.
* 2.RNI testing already planned or performed within the past 12 months.
* 3.Unable to give informed consent.
* 4.Contraindications to or inability to perform exercise treadmill testing or pharmacological testing.
* 5.Medical condition with a prognosis of less than 3.25 years.
* 6.Likely to be unavailable for follow-up.
* 7.Unable to read and understand English or French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2017-03-20 (Estimated); Primary Completion 2021-06-20 (Estimated); Study Completion 2022-06-10 (Estimated)

PRIMARY OUTCOMES:
Combined index (i.e.if any are positive then index is positive) | Yearly up to 3 years from date of randomization
  Myocardial Infarction, Death,Urgent Hospitalization for Cardiac Reasons

SECONDARY OUTCOMES:
Quality of Life | Baseline and yearly up to 3 years from date of randomization
  Difference in scores between baseline and follow-up Seattle Angina Questionnaire

OTHER OUTCOMES:
Resource Utilization | Yearly up to 3 years from date of randomization
  Total number of hospital days for cardiac admissions, further invasive and non-invasive testing, and revascularization procedures

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Joyal, MD, Principal Investigator — Interventional Cardiologist, Assistant Professor of Medicine, McGill University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brindis RG, Douglas PS, Hendel RC, Peterson ED, Wolk MJ, Allen JM, Patel MR, Raskin IE, Hendel RC, Bateman TM, Cerqueira MD, Gibbons RJ, Gillam LD, Gillespie JA, Hendel RC, Iskandrian AE, Jerome SD, Krumholz HM, Messer JV, Spertus JA, Stowers SA; American College of Cardiology Foundation Quality Strategic Directions Committee Appropriateness Criteria Working Group; American Society of Nuclear Cardiology; American Heart Association. ACCF/ASNC appropriateness criteria for single-photon emission computed tomography myocardial perfusion imaging (SPECT MPI): a report of the American College of Cardiology Foundation Quality Strategic Directions Committee Appropriateness Criteria Working Group and the American Society of Nuclear Cardiology endorsed by the American Heart Association. J Am Coll Cardiol. 2005 Oct 18;46(8):1587-605. doi: 10.1016/j.jacc.2005.08.029. PMID 16226194
- [Background] Lloyd-Jones D, Adams RJ, Brown TM, Carnethon M, Dai S, De Simone G, Ferguson TB, Ford E, Furie K, Gillespie C, Go A, Greenlund K, Haase N, Hailpern S, Ho PM, Howard V, Kissela B, Kittner S, Lackland D, Lisabeth L, Marelli A, McDermott MM, Meigs J, Mozaffarian D, Mussolino M, Nichol G, Roger VL, Rosamond W, Sacco R, Sorlie P, Stafford R, Thom T, Wasserthiel-Smoller S, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2010 update: a report from the American Heart Association. Circulation. 2010 Feb 23;121(7):948-54. doi: 10.1161/CIRCULATIONAHA.109.192666. No abstract available. PMID 20177011
- [Background] Hendel RC, Berman DS, Di Carli MF, Heidenreich PA, Henkin RE, Pellikka PA, Pohost GM, Williams KA; American College of Cardiology Foundation Appropriate Use Criteria Task Force; American Society of Nuclear Cardiology; American College of Radiology; American Heart Association; American Society of Echocardiology; Society of Cardiovascular Computed Tomography; Society for Cardiovascular Magnetic Resonance; Society of Nuclear Medicine. ACCF/ASNC/ACR/AHA/ASE/SCCT/SCMR/SNM 2009 Appropriate Use Criteria for Cardiac Radionuclide Imaging: A Report of the American College of Cardiology Foundation Appropriate Use Criteria Task Force, the American Society of Nuclear Cardiology, the American College of Radiology, the American Heart Association, the American Society of Echocardiography, the Society of Cardiovascular Computed Tomography, the Society for Cardiovascular Magnetic Resonance, and the Society of Nuclear Medicine. J Am Coll Cardiol. 2009 Jun 9;53(23):2201-29. doi: 10.1016/j.jacc.2009.02.013. No abstract available. PMID 19497454
- [Background] Fihn SD, Gardin JM, Abrams J, Berra K, Blankenship JC, Dallas AP, Douglas PS, Foody JM, Gerber TC, Hinderliter AL, King SB 3rd, Kligfield PD, Krumholz HM, Kwong RY, Lim MJ, Linderbaum JA, Mack MJ, Munger MA, Prager RL, Sabik JF, Shaw LJ, Sikkema JD, Smith CR Jr, Smith SC Jr, Spertus JA, Williams SV; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines; American College of Physicians; American Association for Thoracic Surgery; Preventive Cardiovascular Nurses Association; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons. 2012 ACCF/AHA/ACP/AATS/PCNA/SCAI/STS Guideline for the diagnosis and management of patients with stable ischemic heart disease: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines, and the American College of Physicians, American Association for Thoracic Surgery, Preventive Cardiovascular Nurses Association, Society for Cardiovascular Angiography and Interventions, and Society of Thoracic Surgeons. J Am Coll Cardiol. 2012 Dec 18;60(24):e44-e164. doi: 10.1016/j.jacc.2012.07.013. Epub 2012 Nov 19. No abstract available. PMID 23182125